CLINICAL TRIAL: NCT03075839
Title: Impact of Switching to Non-Menthol Cigarettes Among Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000020334; 1P50DA036151-01 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Results first posted 2020-04-17 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Within-subject design comparing smoking behavior when using menthol vs. non-menthol cigarettes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cigarette Brand Switching (Experimental): Adult smokers will be switched from using menthol cigarettes to non-menthol cigarettes
  Interventions: Other: Cigarette Brand Switching

INTERVENTIONS:
Other: Cigarette Brand Switching — Adult smokers will be switched from smoking menthol cigarettes to non-menthol cigarettes for a period of two weeks

SUMMARY:
This pilot study will investigate within-person changes in smoking behavior when current adult smokers are systematically switched from smoking menthol cigarettes to non-menthol cigarettes.

DETAILED DESCRIPTION:
The goals of this project include evaluating the feasibility of a cigarette switching paradigm to examine how switching adult smokers from menthol to non-menthol cigarettes impacts smoking behavior and satisfaction. Smoking behavior will be measured by self-reported total number of cigarettes and time to first cigarette in the morning, assessed during the period of menthol smoking (week 1) and again after switching to non-menthol cigarettes (weeks 2, 3). Smoking satisfaction will be measured by self-reported ratings of the cigarettes, assessed during the period of menthol smoking (week 1) and again after switching to non-menthol cigarettes (weeks 2, 3).

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Able to read English
* Cigarette smoker

Exclusion Criteria:

* Seeking smoking cessation treatment
* Serious psychiatric or medical condition
* Use of other drugs
* Unable or unwilling to complete study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krysten Bold, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bold KW, Jatlow P, Fucito LM, Eid T, Krishnan-Sarin S, O'Malley S. Evaluating the effect of switching to non-menthol cigarettes among current menthol smokers: an empirical study of a potential ban of characterising menthol flavour in cigarettes. Tob Control. 2020 Nov;29(6):624-630. doi: 10.1136/tobaccocontrol-2019-055154. Epub 2019 Nov 4. PMID 31685586

RESULTS

PARTICIPANT FLOW:
Groups:
- Cigarette Brand Switching: Adult smokers will be switched from using menthol cigarettes to non-menthol cigarettes
  Cigarette Brand Switching: Adult smokers will be switched from smoking menthol cigarettes to non-menthol cigarettes
Period: Overall Study
Arm/Group | Cigarette Brand Switching
Started | 33
Completed | 29
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Of the 33 participants who were enrolled, four dropped out prior to the intervention phase where they switched from menthol to non-menthol cigarettes, so the final sample for analysis was n=29.
Arm/Group | Cigarette Brand Switching
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 6
  Race/Ethnicity: Non Hispanic Black | 13
  Race/Ethnicity: Non Hispanic White | 11
  Race/Ethnicity: Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Cigarettes Smoked
Description: Change in self-reported total number of cigarettes smoked per day after switching to non-menthol cigarettes
Time Frame: Menthol smoking (Week 2), Non-menthol smoking (Week 4)
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Cigarette Brand Switching
Number analyzed (Participants) | 29
cigarettes per day | 2.2 (3.2)

2. Secondary Outcome: Nicotine Dependence
Description: Self-reported subjective ratings of nicotine dependence after switching to non-menthol cigarettes (measured as change in Wisconsin Inventory of Smoking Dependence Motives (WISDM) total dependence scores). Total range 11-77 with higher scores indicating greater nicotine dependence.
Time Frame: Week 4 (non-menthol)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cigarette Brand Switching
Number analyzed (Participants) | 29
score on a scale | 36.8 (10.9)

3. Secondary Outcome: Quitting Interest
Description: Self-reported subjective motivation/interest in quitting smoking after switching to non-menthol cigarettes. Measured by the item "how important is quitting smoking to you?" from 1 "not at all" to 10 "extremely".
Time Frame: Week 4 (non-menthol)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cigarette Brand Switching
Number analyzed (Participants) | 29
units on a scale | 5.4 (2.5)

ADVERSE EVENTS:
Time Frame: Data were collected while participants were enrolled in the study (duration=4 weeks). Participants were enrolled over a one-year period.
Description: Adverse events were assessed according to clinicaltrials.gov definitions and in accordance with systematic assessment guidelines by the university review board for grading the severity of adverse events.
Arm/Group | Cigarette Brand Switching
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
* Analyses may be under-powered, a larger replication trial is needed
* Some participants continued smoking menthol cigarettes during the study
* Cigarettes were provided to encourage protocol adherence which may impact smoking behavior

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT03075839/Prot_SAP_000.pdf